CLINICAL TRIAL: NCT01401491
Title: Treatment Strategy for Refractory Schizophrenia: Drug Interaction Between Clozapine and Fluvoxamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Mong-Liang Lu, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 95019
Record Dates: First submitted 2011-05-19; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; clozapine; fluvoxamine; metabolic syndrome
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome | interventions — Clozapine; Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- clozapine + fluvoxamine (Active Comparator)
  Interventions: Drug: clozapine plus fluvoxamine
- clozapine + placebo (Placebo Comparator)
  Interventions: Drug: clozapine plus placebo

INTERVENTIONS:
Drug: clozapine plus fluvoxamine — clozapine 100 mg/day plus fluvoxamine 50 mg/day
  Arms: clozapine + fluvoxamine
Drug: clozapine plus placebo — clozapine 300 mg/day plus placebo
  Arms: clozapine + placebo

SUMMARY:
Clozapine has been virtually the only psychopharmacological choice in patients with schizophrenia who either did not response to typical neuroleptics or experienced severe extrapyramidal side effects and consequently did not tolerate this medication. There are patients who do not respond to clozapine, and the need to treat these severely ill patients frequently compels clinicians to adopt therapeutic innovations that lack a sound empirical basis. One strategy is the combination of various other somatic treatments with clozapine.

Recently, the investigators conduct a preliminary open trial to evaluate the safety and efficacy of fluvoxamine coadministration with clozapine in refractory schizophrenic patients. The combined treatment is well tolerated, and clinical improvement is observed in our patients. And the concomitant fluvoxamine could attenuate the clozapine-induced weight gain and metabolic disturbance. However, the effects of fluvoxamine on the safety and therapeutic efficacy of clozapine need to be further clarified in double-blind study.

DETAILED DESCRIPTION:
Background Schizophrenia is one of the most severe mental illnesses. The prevalence of schizophrenia has been variously reported as ranging from 1 to 1.5 percent. More than 50% of patients can be described as having a poor outcome, with repeated hospitalizations, exacerbations of symptoms, episodes of major mood disorders, and suicide attempts. Schizophrenia is costly in medical care, treatment and rehabilitation, and reduced or lost productivity. Therefore, the development of effective treatment for schizophrenic patients is an important issue.

The classical antipsychotic drugs are the dopamine receptor antagonists, which are effective in the treatment of schizophrenia, particularly of the positive symptoms. Even with treatment of typical antipsychotics, about 50% of schizophrenic patients lead severely debilitated lives. Second, the classical antipsychotic drugs are associated with annoying and serious adverse effects. Clozapine has been virtually the only psychopharmacological choice in patients with schizophrenia who either did not response to typical neuroleptics or experienced severe extrapyramidal side effects and consequently did not tolerate this medication. There are patients who do not respond to clozapine, and the need to treat these severely ill patients frequently compels clinicians to adopt therapeutic innovations that lack a sound empirical basis. One strategy is the combination of various other somatic treatments with clozapine.

Recently, the investigators conduct a preliminary open trial to evaluate the safety and efficacy of fluvoxamine coadministration with clozapine in refractory schizophrenic patients. The mean plasma clozapine levels obtained by clozapine 100 mg/day plus fluvoxamine 50 mg/day is close to that produced by 300-mg/day clozapine monotherapy in one of our previous studies. The combined treatment is well tolerated, and clinical improvement is observed in our patients. And the concomitant fluvoxamine could attenuate the clozapine-induced weight gain and metabolic disturbance. However, the effects of fluvoxamine on the safety and therapeutic efficacy of clozapine need to be further clarified in double-blind study.

Methods This study is a three-year proposal. Sixty treatment-resistant schizophrenic inpatients will participate in this project. The subjects will be randomized to one of two parallel groups: clozapine monotherapy and clozapine plus fluvoxamine treatment. The double-blind active treatment will consist of two periods.

The measures of clinical efficacy will be the Positive And Negative Syndrome Scale, Clinical Global Impression, and Nurses'Observation Scale for Inpatient Evaluation. The measures of side effects will be the Extrapyramidal Symptom Rating Scale and the UKU Side Effect Rating Scale. Fasting serum samples are collected to determine the lipid profile (total cholesterol, triglycerides, HDL, and LDL), glucose level, and insulin level. Plasma levels of clozapine, norclozapine, and clozapine N-oxide will be determined by high performance liquid chromatography with ultraviolet detection.

The following results are expected:

1. In treatment-resistant schizophrenic patients, global antipsychotic effect of clozapine plus fluvoxamine treatment is superior to clozapine monotherapy.
2. Clozapine plus fluvoxamine treatment has less adverse effects than clozapine monotherapy.
3. The effect of clozapine plus fluvoxamine treatment on body weight and metabolic disturbances is superior to clozapine monotherapy.
4. Steady-state plasma levels of clozapine and its metabolites account for a proportion of variance of clinical effects.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients meet the DSM-IV criteria for schizophrenia.
2. Treatment refractoriness: Failed to respond to at least two typical neuroleptics at dosage equivalent to or greater than 1000 mg/day of chlorpromazine for a period of at least six weeks.
3. Age 18-60 years.
4. Males or females.
5. Total PANSS score >60
6. Good physical health determined by complete physical examination, laboratory tests, and EKG.
7. Capacity and willingness to give written informed consent.

Exclusion Criteria:

1. History of illicit substance abuse or dependence
2. History of clozapine intolerance (such as clinically significant leukopenia or agranulocytosis).
3. Patients with WBC count less than 3500/mm3 or ANC count less than 2000/mm3will not be included.
4. Any depot neuroleptics within 30 days before the day of randomization.
5. Epilepsy, active hepatitis, HIV positivity, or current myeloproliferative disorder. Other medical illnesses may necessitate subjects' exclusion after evaluation of individual cases by the principal investigator and other staffs. Clinical judgment will be used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
the changes in the psychopathology during the trial | every 2 weeks
  The changes in the scores of psychopathology assessment (the Positive and Negative Syndrome Scale, PANSS)
the changes in the metabolic syndrome parameters during the trial | every 2 weeks
  The changes in the metabolic syndrome parameters

SECONDARY OUTCOMES:
the changes in the plasma drug levels | every 2 weeks
  the plasma levels of fluvoxamine, clozapine, and its metabolites
The changes in insulin levels | every 2 weeks
  The changes in insulin levels
The changes in the depression severity | every 2 weeks
  The changes in the scores of the Hamilton Rating Scale for Depression
The changes in the adipokine levels | every 2 weeks
  The changes in the adipokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Mong-Liang Lu, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lu ML, Chen TT, Kuo PH, Hsu CC, Chen CH. Effects of adjunctive fluvoxamine on metabolic parameters and psychopathology in clozapine-treated patients with schizophrenia: A 12-week, randomized, double-blind, placebo-controlled study. Schizophr Res. 2018 Mar;193:126-133. doi: 10.1016/j.schres.2017.06.030. Epub 2017 Jul 6. PMID 28688742